CLINICAL TRIAL: NCT00113607
Title: An Open-Label Multicenter Randomized Phase 3 Study Comparing the Combination of DOXIL/CAELYX and YONDELIS With DOXIL/CAELYX Alone in Subjects With Advanced Relapsed Ovarian Cancer
Brief Title: An Efficacy and Safety Study for Yondelis (Trabectedin) in Patients With Advanced Relapsed Ovarian Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR003448; ET743-OVA-301 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.); 2004-005276-16 (EudraCT Number)
Record Dates: First submitted 2005-06-09; First posted 2005-06-10 (Estimated); Results first posted 2013-08-23 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer; Trabectedin; Yondelis; Advanced Relapsed Ovarian Cancer; DOXIL; CAELYX
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Trabectedin; liposomal doxorubicin; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DOXIL + trabectedin (Experimental): Combination arm - Trabectedin + DOXIL: DOXIL 30 mg/m2 intravenous (IV) infusion over 90 minutes + trabectedin 1.1 mg/m2 IV infusion over 3 hours every 3 weeks. patients will be premedicated with 20 mg dexamethasone or its equivalent IV infusion over 30 minutes prior to the DOXIL infusion.
  Interventions: Drug: Trabectedin; Drug: DOXIL; Drug: Dexamethasone
- DOXIL (Active Comparator): Monotherapy arm - DOXIL: 50 mg/m2 IV infusion over 90 minutes every 4 weeks.
  Interventions: Drug: DOXIL

INTERVENTIONS:
Drug: Trabectedin — Type=exact number, unit=mg/m2, number=1.1, form=solution, route=IV. Trabectedin will be administered over 3 hours every 3 weeks.
  Other Names: Yondelis
  Arms: DOXIL + trabectedin
Drug: DOXIL — Type=exact number, unit=mg/m2, number=30, 50, form=solution, route=IV. DOXIL will be administered over 90 minutes every 4 weeks when administered alone (monotherapy) and every 3 weeks when administered with trabectedin.
  Other Names: CAELYX
Drug: Dexamethasone — Type=exact number, unit=mg, number=20, form=solution, route=IV. Dexamethasone or its equivalent will be administered over 30 minutes prior to the DOXIL infusion.
  Arms: DOXIL + trabectedin

SUMMARY:
The purpose of the study is to compare the progression-free survival (PFS) of the combination of trabectedin + DOXIL with DOXIL monotherapy in patients with ovarian cancer.

DETAILED DESCRIPTION:
This is a multicenter, open-label (all people know the identity of the intervention), randomized (study medication is assigned by chance), Phase 3 study comparing the combination of trabectedin + DOXIL with DOXIL monotherapy in patients with advanced ovarian cancer (who were previously treated and for whom first-line platinum-based chemotherapy regimen has failed). Approximately 650 patients will be randomly assigned to 1 of the treatment arms (DOXIL and DOXIL + trabectedin) over 2 years. At the time of randomization, patients will be stratified on the basis of platinum sensitivity of disease (sensitive or resistant) and baseline Eastern Cooperative Oncology Group performance status score (0 to 1 or 2. Safety will be evaluated on the basis of adverse events, clinical laboratory tests, physical examination, vital signs assessment and cardiovascular safety assessment. An interim analysis of overall survival will be performed in conjunction with progression-free survival analysis during the study. Treatment will be continued until disease progression occurred or until patients experienced a confirmed complete response for at least 2 cycles. Continuation of treatment in select individual patients beyond this study end date will be allowed if the investigator determined that the patient is benefiting from treatment, is eligible to receive further therapy, and consents to treatment. If disease progression has not occurred at treatment termination, then disease assessment will continue every 8 weeks until there is evidence of disease progression or death, or until the clinical data cutoff date, or until the start of first subsequent anticancer therapy, whichever is earlier.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven epithelial ovarian cancer, epithelial fallopian tube cancer, or primary peritoneal cancer
* Prior treatment with only 1 platinum based chemotherapy regimen
* Eastern Cooperative Oncology Group status of not more than 2
* Progression more than 6 months after the start of initial chemotherapy treatment

Exclusion Criteria:

* Treatment with more than 1 prior chemotherapy regimen
* Progression within 6 months after starting initial chemotherapy
* Prior exposure to anthracyclines
* Unwilling or unable to have central venous catheter
* Known clinically relevant central nervous system metastasis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 672 (Actual)
Dates: Start 2005-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (111):
- United States (28):
  - Mobile, Alabama
  - Tucson, Arizona
  - Los Angeles, California
  - Newport Beach, California
  - Orange, California
  - Englewood, Colorado
  - Stamford, Connecticut
  - Tampa, Florida
  - Coeur d'Alene, Idaho
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Morristown, New Jersey
  - New York, New York
  - Charlotte, North Carolina
  - Greenville, North Carolina
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Toledo, Ohio
  - Portland, Oregon
  - Pittsburgh, Pennsylvania
  - Greenville, South Carolina
  - Chattanooga, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - Galveston, Texas
- Argentina (3):
  - Buenos Aires
  - Mendoza
  - Sante Fe
- Australia (5):
  - Adelaide
  - Bentleigh
  - Douglas
  - St Leonards
  - Toorak Gardens
- Belgium (4):
  - Edegem
  - Hasselt
  - Leuven
  - Wilrijk
- Brazil (6):
  - Barretos
  - Belo Horizonte
  - Cerqueira César
  - Londrina
  - Santo André
  - São Paulo
- Canada (5):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Ottawa, Ontario
  - Montreal, Quebec
  - Québec, Quebec
- Chile (2):
  - Reneca
  - Santiago
- China (5):
  - Beijing
  - Guangzhou
  - Hangzhou
  - Jinan
  - Shanghai
- France (3):
  - Chartres
  - Paris
  - Pierre-Bénite
- Germany (7):
  - Düsseldorf
  - Heidelberg
  - Jena
  - Karlsruhe
  - Mainz
  - Villingen-Schwenningen
  - Wilhelmshaven
- Hong Kong (3):
  - Chai Wan
  - Hong Kong
  - Shatin
- Netherlands (4):
  - Amsterdam
  - Enschede
  - Groningen
  - Maastricht
- Poland (7):
  - Gdansku
  - Gliwice
  - Krakow
  - Olsztyn
  - Poznan
  - Warszawa Poland
  - Wroclaw
- Russia (6):
  - Chelyabinsk
  - Moscow
  - Obninsk, Kaluga Region
  - Orenburg
  - Saint Petersburg
  - Samara
- Singapore, Singapore
- Seoul, South Korea
- Spain (8):
  - Barcelona
  - Girona
  - Guadalajara
  - L'Hospitalet de Llobregat
  - Madrid
  - Marañón
  - Valencia
  - Zaragoza
- Sweden (3):
  - Gothenburg
  - Umeå
  - Uppsala
- Taiwan (3):
  - Kaohsiung County
  - Taipei
  - Taoyuan District
- United Kingdom (7):
  - Birmingham
  - Edinburgh
  - Leicester
  - London
  - Nottingham
  - Poole
  - Sheffield

REFERENCES:
- [Derived] Newhouse R, Nelissen E, El-Shakankery KH, Rogozinska E, Bain E, Veiga S, Morrison J. Pegylated liposomal doxorubicin for relapsed epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Jul 5;7(7):CD006910. doi: 10.1002/14651858.CD006910.pub3. PMID 37407274
- [Derived] Jones RL, Herzog TJ, Patel SR, von Mehren M, Schuetze SM, Van Tine BA, Coleman RL, Knoblauch R, Triantos S, Hu P, Shalaby W, McGowan T, Monk BJ, Demetri GD. Cardiac safety of trabectedin monotherapy or in combination with pegylated liposomal doxorubicin in patients with sarcomas and ovarian cancer. Cancer Med. 2021 Jun;10(11):3565-3574. doi: 10.1002/cam4.3903. Epub 2021 May 7. PMID 33960681
- [Derived] Krasner CN, Poveda A, Herzog TJ, Vermorken JB, Kaye SB, Nieto A, Claret PL, Park YC, Parekh T, Monk BJ. Patient-reported outcomes in relapsed ovarian cancer: results from a randomized Phase III study of trabectedin with pegylated liposomal doxorubicin (PLD) versus PLD alone. Gynecol Oncol. 2012 Oct;127(1):161-7. doi: 10.1016/j.ygyno.2012.06.034. Epub 2012 Jul 2. PMID 22765965
- [Derived] Monk BJ, Herzog TJ, Kaye SB, Krasner CN, Vermorken JB, Muggia FM, Pujade-Lauraine E, Park YC, Parekh TV, Poveda AM. Trabectedin plus pegylated liposomal doxorubicin (PLD) versus PLD in recurrent ovarian cancer: overall survival analysis. Eur J Cancer. 2012 Oct;48(15):2361-8. doi: 10.1016/j.ejca.2012.04.001. Epub 2012 Apr 26. PMID 22541893
- See also: Monk BJ, Herzog TJ, Kaye SB, Krasner CN, Vermorken JB, Muggia FM, Pujade-Lauraine E, Lisyanskaya AS, Makhson AN, Rolski J, Gorbounova VA, Ghatage P, Bidzinski M, Shen K, Ngan HY, Vergote IB, Nam JH, Park YC, Lebedinsky CA, Poveda AM. — http://www.ncbi.nlm.nih.gov/pubmed/20516432
- See also: Monk BJ, Herzog TJ, Kaye SB, Krasner CN, Vermorken JB, Muggia FM, Pujade-Lauraine E, Park YC, Parekh TV, Poveda AM. Trabectedin plus pegylated liposomal doxorubicin (PLD) versus PLD in recurrent ovarian cancer: Overall survival analysis. — http://www.ncbi.nlm.nih.gov/pubmed/22541893

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in a total of 21 countries at 124 sites worldwide.
Pre-assignment Details: 672 participants were randomized (337 in trabectedin + DOXIL arm and 335 in DOXIL arm) and out of which 9 participants were not treated. 663 participants received treatment ie, 330 participants received DOXIL and 333 received trabectedin + DOXIL.
Groups:
- DOXIL: 50 mg/m2 DOXIL administered as a 90-minute intravenous (IV) infusion, every 4 weeks
- Trabectedin/DOXIL: 30 mg/m2 DOXIL administered as a 90-minute IV infusion followed by 1.1 mg/m2 trabectedin as a 3-hour IV infusion, every 3 weeks
Period: Overall Study
Arm/Group | DOXIL | Trabectedin/DOXIL
Started | 335 (Number of randomized participants) | 337 (Number of randomized participants)
Completed | 0 | 0
Not Completed | 335 | 337
Not completed — Adverse Event | 40 | 71
Not completed — Death | 8 | 8
Not completed — Withdrawal by Subject | 50 | 58
Not completed — Lost to Follow-up | 0 | 2
Not completed — Disease Progression | 180 | 142
Not completed — Complete Response (Confirmed) | 14 | 24
Not completed — Other | 43 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DOXIL | Trabectedin/DOXIL | Total
Number analyzed (Participants) | 335 | 337 | 672
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (10.75) | 56.8 (10.48) | 57.5 (10.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 335 | 337 | 672
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Argentina | 5 | 2 | 7
  Australia | 5 | 2 | 7
  Belgium-Luxemburg | 12 | 13 | 25
  Brazil | 12 | 9 | 21
  Canada | 22 | 34 | 56
  Chile | 1 | 2 | 3
  France | 0 | 2 | 2
  Germany | 6 | 13 | 19
  Hong Kong | 10 | 15 | 25
  Italy | 3 | 4 | 7
  Netherlands | 4 | 1 | 5
  China | 37 | 36 | 73
  Poland | 47 | 39 | 86
  Republic Of Korea | 17 | 11 | 28
  Russia | 52 | 56 | 108
  Singapore | 0 | 1 | 1
  Spain | 8 | 9 | 17
  Sweden | 6 | 8 | 14
  Taiwan | 7 | 2 | 9
  United Kingdom | 18 | 20 | 38
  United States Of America | 63 | 58 | 121

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS): Independent Radiologist Review
Description: PFS is defined as the time between randomization and disease progression or death.
Time Frame: From the date of randomization until the date of disease progression or death, as assessed for approximately 3 years
Population: All Measurable Analysis Participants: All randomized participants who had measurable disease at baseline as assessed by the independent radiology review. Measurable disease is defined as having at least 1 lesion measured with a diameter of ≥20 mm using conventional techniques or of ≥10 mm using a spiral computerized tomography scan.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | DOXIL | Trabectedin/DOXIL
Number analyzed (Participants) | 317 | 328
Months | 5.8 [5.5 to 7.1] | 7.3 [5.9 to 7.9]
Statistical Analysis 1: Comparison: DOXIL vs Trabectedin/DOXIL; Test type: Superiority or Other; p = 0.0190, Log Rank; Hazard Ratio, log = 0.79, 95% CI 2-sided [0.65 to 0.96]

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time between the randomization and death
Time Frame: From the date of randomization until the date of death, as assessed for approximately 3 years
Population: All Randomized Analysis Participants: all participants who were randomized to this study, independent of whether they received study medication or not
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | DOXIL | Trabectedin/DOXIL
Number analyzed (Participants) | 335 | 337
Months | 18.9 [17.1 to 21.5] | 22.2 [19.3 to 25.0]
Statistical Analysis 1: Comparison: DOXIL vs Trabectedin/DOXIL; Test type: Superiority or Other; p = 0.0835, Log Rank; Hazard Ratio, log = 0.86, 95% CI 2-sided [0.72 to 1.02]

3. Secondary Outcome: Objective Response Rate (ORR) - Independent Radiologist Review
Description: Percentage of participants who achieved complete response (CR) or partial response (PR) as best overall response. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR) = Disappearance of all target lesions; Partial Response (PR)= greater than or equal to 30% decrease in the sum of the longest diameter of target lesions and Overall Response (OR) = CR + PR.
Time Frame: From the date of randomization until the date of disease progression or death, as assessed for approximately 3 years
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | DOXIL | Trabectedin/DOXIL
Number analyzed (Participants) | 335 | 337
Percentage of participants | 18.8 | 27.6
Statistical Analysis 1: Comparison: DOXIL vs Trabectedin/DOXIL; Test type: Superiority or Other; p = 0.0080, Fisher Exact; Odds Ratio (OR) = 1.646, 95% CI 2-sided [1.144 to 2.367]

4. Secondary Outcome: Duration of Response: Independent Radiologist Review
Description: Duration of response was defined only for participants who had complete response or partial response as best overall response. Duration of response was calculated from the date of first documentation of response (not the confirmation) to the date of disease progression or death due to progressive disease.
Time Frame: From the date of first documentation of response to the date of disease progression or death due to progressive disease, as assessed for approximately 3 years
Population: All Responders (CR/PR) Analysis Participants: all participants who achieved CR or PR as best overall response during the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | DOXIL | Trabectedin/DOXIL
Number analyzed (Participants) | 63 | 93
Months | 7.7 [6.5 to 9.0] | 7.9 [7.4 to 9.2]
Statistical Analysis 1: Comparison: DOXIL vs Trabectedin/DOXIL; Test type: Superiority or Other; p = 0.8203, Log Rank; Hazard Ratio, log = 0.95, 95% CI 2-sided [0.62 to 1.46]

5. Secondary Outcome: Median Area Under Curve (AUC) of Trabectedin.
Description: Median simulated area under the curve (AUC) of a 21 day trabectedin profile of participants (of this study) administering trabectedin and doxil, calculated using the trapezoidal rule method. Simulations were based on a dataset created of 1000 participants using the posthoc parameter estimations, derived from the population pharmacokinetic analysis dataset of Trabectedin (Participants=831, with resampling). Plasma concentration-time profiles were simulated up to 504 hour post-dosing using a rich sampling.
Time Frame: Day 1 (Predose; 1.5 hour after start of infusion; 5 minutes, 2 hour and 6 to 20 hour after end of infusion); Day 8 (168 hour after end of infusion); and Day 15 (336 hour after end of infusion) at Cycles 1 and 2
Population: Blood samples for pharmacokinetic analysis were collected from 86 participants of this study.
Measure: Number; unit: ng*h/mL
Arm/Group | Trabectedin/DOXIL
Number analyzed (Participants) | 86
ng*h/mL | 74.24

6. Secondary Outcome: Median Maximum Plasma Concentration (Cmax) of Trabectedin.
Description: Median simulated maximum plasma concentration (Cmax) at 3 hour of a 21 day trabectedin profile of participants (of this study) administering trabectedin and doxil. The assessment of Cmax was based on a dataset created of 1000 participants using the posthoc parameter estimations, derived from the population pharmacokinetic analysis dataset of Trabectedin (participants=831, with resampling). Plasma concentration-time profiles were simulated up to 504 hour post-dosing using a rich sampling.
Time Frame: as for outcome 5
Population: Blood samples for pharmacokinetic analysis were collected from 86 participants of this study.
Measure: Number; unit: pg/mL
Arm/Group | Trabectedin/DOXIL
Number analyzed (Participants) | 86
pg/mL | 13394

ADVERSE EVENTS:
Time Frame: From the time of the first study-related procedure until up to 30 days after administration of the last dose of study medication.
Description: Number of treated participants were analyzed for adverse events. 672 participants were randomized (337 in trabectedin + DOXIL arm and 335 in DOXIL arm), out of which 663 participants received treatment ie, 330 participants received DOXIL and 333 received trabectedin + DOXIL and were analyzed for adverse events.
Arm/Group | Trabectedin/DOXIL | DOXIL
Serious Adverse Events (participants affected / at risk) | 133/333 | 102/330
Other Adverse Events (participants affected / at risk) | 333/333 | 318/330
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trabectedin/DOXIL (N=333) | DOXIL (N=330)
Anaemia (Blood and lymphatic system disorders) | 17 | 7
Bicytopenia (Blood and lymphatic system disorders) | 1 | 0
Bone Marrow Failure (Blood and lymphatic system disorders) | 4 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 18 | 5
Granulocytopenia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 16 | 3
Neutropenia (Blood and lymphatic system disorders) | 26 | 7
Pancytopenia (Blood and lymphatic system disorders) | 6 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 21 | 1
Cardiac Arrest (Cardiac disorders) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 2 | 1
Electromechanical Dissociation (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Ventricular Tachycardia (Cardiac disorders) | 1 | 0
Adenomatous Polyposis Coli (Congenital, familial and genetic disorders) | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 3 | 1
Abdominal Pain (Gastrointestinal disorders) | 6 | 9
Aphthous Stomatitis (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 6 | 7
Colonic Obstruction (Gastrointestinal disorders) | 3 | 2
Constipation (Gastrointestinal disorders) | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 6 | 3
Enterocutaneous Fistula (Gastrointestinal disorders) | 1 | 0
Erosive Oesophagitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Obstruction (Gastrointestinal disorders) | 0 | 2
Ileus (Gastrointestinal disorders) | 1 | 4
Intestinal Fistula (Gastrointestinal disorders) | 1 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 7 | 11
Large Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Mechanical Ileus (Gastrointestinal disorders) | 0 | 2
Mouth Ulceration (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 14 | 8
Oesophageal Ulcer (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 2
Small Intestinal Obstruction (Gastrointestinal disorders) | 7 | 3
Stomatitis (Gastrointestinal disorders) | 1 | 2
Subileus (Gastrointestinal disorders) | 1 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 15 | 8
Adverse Drug Reaction (General disorders) | 1 | 1
Asthenia (General disorders) | 0 | 2
Catheter Related Complication (General disorders) | 2 | 0
Catheter Site Phlebitis (General disorders) | 1 | 0
Chest Discomfort (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Condition Aggravated (General disorders) | 1 | 0
Extravasation (General disorders) | 1 | 0
Fatigue (General disorders) | 8 | 1
General Physical Health Deterioration (General disorders) | 3 | 3
Hernia Obstructive (General disorders) | 0 | 1
Hernia Pain (General disorders) | 1 | 0
Mucosal Inflammation (General disorders) | 0 | 3
Non-Cardiac Chest Pain (General disorders) | 2 | 1
Oedema Peripheral (General disorders) | 3 | 0
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 10 | 3
Sudden Death (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatitis Cholestatic (Hepatobiliary disorders) | 0 | 1
Hepatitis Toxic (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0
Anaphylactic Reaction (Immune system disorders) | 0 | 2
Drug Hypersensitivity (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 2 | 3
Abscess (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 3 | 0
Bacterial Sepsis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Catheter Related Infection (Infections and infestations) | 3 | 1
Catheter Sepsis (Infections and infestations) | 1 | 0
Catheter Site Cellulitis (Infections and infestations) | 0 | 1
Catheter Site Infection (Infections and infestations) | 4 | 0
Cellulitis (Infections and infestations) | 1 | 1
Central Line Infection (Infections and infestations) | 1 | 0
Clostridium Difficile Colitis (Infections and infestations) | 1 | 0
Enterocolitis Infectious (Infections and infestations) | 0 | 1
Erysipeloid (Infections and infestations) | 0 | 1
Helicobacter Gastritis (Infections and infestations) | 1 | 0
Herpes Oesophagitis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 2
Influenza (Infections and infestations) | 1 | 0
Neutropenic Infection (Infections and infestations) | 3 | 0
Neutropenic Sepsis (Infections and infestations) | 2 | 0
Oesophageal Candidiasis (Infections and infestations) | 0 | 1
Perineal Abscess (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 4
Pyelonephritis (Infections and infestations) | 0 | 1
Respiratory Tract Infection Viral (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 2
Septic Shock (Infections and infestations) | 1 | 0
Staphylococcal Sepsis (Infections and infestations) | 1 | 0
Subcutaneous Abscess (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 2 | 2
Urinary Tract Infection Bacterial (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Device Dislocation (Injury, poisoning and procedural complications) | 0 | 1
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1
Medical Device Complication (Injury, poisoning and procedural complications) | 1 | 0
Postoperative Ileus (Injury, poisoning and procedural complications) | 1 | 0
Procedural Nausea (Injury, poisoning and procedural complications) | 0 | 1
Procedural Vomiting (Injury, poisoning and procedural complications) | 0 | 1
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 5 | 0
Aspartate Aminotransferase Increased (Investigations) | 5 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 3 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 1 | 0
Blood Creatinine Increased (Investigations) | 1 | 0
Carbohydrate Antigen 125 Increased (Investigations) | 1 | 0
Electrocardiogram Change (Investigations) | 1 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 1 | 0
Hepatic Enzyme Increased (Investigations) | 1 | 0
Liver Function Test Abnormal (Investigations) | 1 | 0
Transaminases Increased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 3 | 6
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 7 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to Soft Tissue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oncologic Complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Paraneoplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Grand Mal Convulsion (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 2
Loss of Consciousness (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Syncope Vasovagal (Nervous system disorders) | 1 | 0
Confusional State (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Obstructive Uropathy (Renal and urinary disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 3 | 2
Renal Impairment (Renal and urinary disorders) | 1 | 0
Oedema Genital (Reproductive system and breast disorders) | 1 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 13 | 6
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Melanosis (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Arterial Insufficiency (Vascular disorders) | 1 | 0
Axillary Vein Thrombosis (Vascular disorders) | 2 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 2
Haemorrhage (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Jugular Vein Thrombosis (Vascular disorders) | 1 | 0
Peripheral Ischaemia (Vascular disorders) | 1 | 0
Subclavian Vein Thrombosis (Vascular disorders) | 2 | 0
Thrombosis (Vascular disorders) | 3 | 0
Vena Cava Thrombosis (Vascular disorders) | 0 | 1
Venous Occlusion (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trabectedin/DOXIL (N=333) | DOXIL (N=330)
Anaemia (Blood and lymphatic system disorders) | 160 | 82
Leukopenia (Blood and lymphatic system disorders) | 164 | 91
Neutropenia (Blood and lymphatic system disorders) | 256 | 128
Thrombocytopenia (Blood and lymphatic system disorders) | 115 | 27
Abdominal Distension (Gastrointestinal disorders) | 18 | 23
Abdominal Pain (Gastrointestinal disorders) | 70 | 76
Abdominal Pain Upper (Gastrointestinal disorders) | 19 | 25
Ascites (Gastrointestinal disorders) | 13 | 18
Constipation (Gastrointestinal disorders) | 109 | 92
Diarrhoea (Gastrointestinal disorders) | 84 | 63
Dyspepsia (Gastrointestinal disorders) | 43 | 35
Mouth Ulceration (Gastrointestinal disorders) | 11 | 21
Nausea (Gastrointestinal disorders) | 251 | 139
Stomatitis (Gastrointestinal disorders) | 67 | 108
Vomiting (Gastrointestinal disorders) | 188 | 97
Asthenia (General disorders) | 56 | 38
Fatigue (General disorders) | 153 | 122
Mucosal Inflammation (General disorders) | 42 | 64
Oedema Peripheral (General disorders) | 30 | 28
Pain (General disorders) | 18 | 12
Pyrexia (General disorders) | 63 | 44
Hyperbilirubinaemia (Hepatobiliary disorders) | 51 | 25
Urinary Tract Infection (Infections and infestations) | 15 | 19
Alanine Aminotransferase Increased (Investigations) | 185 | 33
Aspartate Aminotransferase Increased (Investigations) | 139 | 35
Blood Alkaline Phosphatase Increased (Investigations) | 77 | 29
Blood Creatine Phosphokinase Increased (Investigations) | 23 | 11
Blood Creatinine Increased (Investigations) | 21 | 20
Anorexia (Metabolism and nutrition disorders) | 109 | 85
Hypoalbuminaemia (Metabolism and nutrition disorders) | 22 | 19
Hypokalaemia (Metabolism and nutrition disorders) | 38 | 26
Hyponatraemia (Metabolism and nutrition disorders) | 19 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 14
Back Pain (Musculoskeletal and connective tissue disorders) | 30 | 31
Myalgia (Musculoskeletal and connective tissue disorders) | 18 | 12
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 20 | 18
Dizziness (Nervous system disorders) | 33 | 22
Dysgeusia (Nervous system disorders) | 19 | 10
Headache (Nervous system disorders) | 55 | 24
Anxiety (Psychiatric disorders) | 23 | 11
Insomnia (Psychiatric disorders) | 34 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 41 | 40
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 52 | 33
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 17 | 24
Alopecia (Skin and subcutaneous tissue disorders) | 42 | 48
Dry Skin (Skin and subcutaneous tissue disorders) | 18 | 10
Erythema (Skin and subcutaneous tissue disorders) | 18 | 19
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 86 | 179
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 20
Rash (Skin and subcutaneous tissue disorders) | 36 | 59
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 21 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days